CLINICAL TRIAL: NCT05751681
Title: Dydrogesterone-Primed Ovarian Stimulation Protocol Versus Gonadotropin Releasing Hormone Antagonist Protocol in Patients With Polycystic Ovary Syndrome Undergoing Intra-Cytoplasmic Sperm Injection
Brief Title: Dydrogesterone-Primed Ovarian Stimulation Protocol Versus Gonadotropin Releasing Hormone Antagonist Protocol in ICSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9736-20-9-2022
Record Dates: First submitted 2022-12-14; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Ovary Cyst; Fertility Issues
Keywords: IVF,ICSI,success rate
MeSH Terms: conditions — Ovarian Cysts; Infertility | interventions — Dydrogesterone; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): will be subjected to progestin primed ovarian stimulation protocol Women in group (A), will be prescribed 20 mg oral dose of dydrogesterone (Duphaston, Abbott) from the 2nd day of the cycle and continued until the trigger day. Transvaginal follicular monitoring will be done for all patients starting the 6th day of cycle.
  Interventions: Other: progestin primed ovarian stimulation protocol; Drug: dydrogesterone (Duphaston, Abbott)
- group (B) (Active Comparator): Gonadotropin Releasing Hormone Antagonist Protocol when the size of dominant follicles reaches 12-13 mm, 0.25 mg of cetrotide (Merck-Serono Germany) will be injected subcutaneously daily and continued until the day of trigger shot.
  Interventions: Other: progestin primed ovarian stimulation protocol; Drug: Cetrotide

INTERVENTIONS:
Other: progestin primed ovarian stimulation protocol — progestin primed ovarian stimulation protocol
Drug: dydrogesterone (Duphaston, Abbott) — 20 mg oral dose of dydrogesterone (Duphaston, Abbott)
  Arms: Group (A)
Drug: Cetrotide — 0.25 mg of Cetrotide (gonadotropin releasing hormone (GnRH) antagonist)
  Other Names: cetrorelix
  Arms: group (B)

SUMMARY:
GnRH antagonist protocol is currently a good strategy for controlled ovarian stimulation in women with PCOS undergoing IVF/ICSI cycles. Finding a protocol that can be a better alternative will help in improving the success rate of IVF/ICSI cycles

DETAILED DESCRIPTION:
Progesterone has potent restraint on hypothalamus-pituitary-ovarian axis. It acts on unidentified hypothalamic pulse oscillator neurons. In turn, it acts on gonadotropins releasing hormone (GnRH) secreting neurons leading to inhibition of GnRH secretion. This results in inhibition of both luteinizing hormone (LH) and follicle-stimulating hormone (FSH) secretion from anterior pituitary. The effect of progesterone appears to decrease GnRH pulse frequency which results in slowing down LH pulse frequency and reducing LH plasma concentrations

ELIGIBILITY:
Inclusion Criteria:

1. All patients should be candidates for ICSI.
2. Age between 20-40 years.
3. Body mass index 18-35 kg/m2.
4. Diagnosis of PCOS according to modified Rotterdam's criteria

Exclusion Criteria:

* 1) Any patient with contraindication to IVF treatment or pregnancy 2) Women with history of intra-uterine abnormality. 3) Severe endometriosis (grade 3 or 4) 4) Clinically significant systemic disease or other endocrinopathy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 20-40 years
Enrollment: 79 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy (Number of MII oocytes retrieved) | 3 months
  this outcome means to measure Percentage (number) of MII oocytes retrieved During our study
Efficacy (Maturation index) | 3 months
  Maturation index will be calculated: Rate of metaphase-II oocytes (MII) to total oocytes

CONTACTS AND LOCATIONS:
Overall Officials: mostafa fahmy, mcs, Principal Investigator — zagazig
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No